CLINICAL TRIAL: NCT06970379
Title: Comparison Between T-prf Versus T-prf and Low-level Laser Stimulation on Bone Healing at Posterior Mandibular Fractures (Randomized Clinical Trial)
Brief Title: T-prf Versus T-prf and Low-level Laser Stimulation on Bone Healing at Posterior Mandibular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0855-02/2024
Record Dates: First submitted 2025-05-13; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Posterior Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T-PRF (Experimental)
  Interventions: Other: T-PRF
- T-PRF and LLLT (Experimental)
  Interventions: Other: T-PRF and Laser biomodulation

INTERVENTIONS:
Other: T-PRF — Patients received T-PRF placement at the fracture line.
  Arms: T-PRF
Other: T-PRF and Laser biomodulation — Subjects underwent the process of bio-stimulation of the fracture line using low-level laser therapy. Wavelength [λ]: 660 nm, Power: 100 mW, Spot size [Ø]: 0.06 cm2, and for 60 seconds
  Arms: T-PRF and LLLT

SUMMARY:
Different types of grafting substances have been used in the recent decade to accelerate bone healing at large bony facial defects. PRF was one of the gold standard materials to be used until it was replaced by its successor T-PRF due to the PRF hazards of preparation. However, T-PRF- still can't stand alone in full bone enhancement procedure. Therefore, the combination with another bone bio-modulation technique, like Low-level Laser Therapy, is a must to approach the full advantage of bone healing. Aim: To compare between the effect of using T-PRF versus T-PRF with Low Level Laser stimulation on bone healing at posterior mandibular fractures

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from posterior mandibular fracture

Exclusion Criteria:

* Patients with an untreated old Mandibular fracture.
* Patient with hematological diseases (thrombocytopenia, hemorrhagic disease, and diabetes).
* Comminuted fracture with bone loss.
* There is an infection at the fracture line.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Change in bone density | Baseline and 3 months
  immediate postoperative CT-scan will be performed and compared with another CT-scan done 12 weeks (3 months) later. The on-demand software (OnDemand 3D APP-DBM, Cybermed, Seoul, South Korea) will be used to calculate bone mineral density in Hounsfield Units (HU). Six measurements will be taken along the fracture line, and the mean will be measured for each patient.
Change in mouth opening | baseline, 24 hrs, 1 week, 4 weeks, 6 weeks, 12 weeks
  With the help of a millimeter ruler, the maximal inter-incisal distance is going to be assessed
Change in wound healing | baseline, 24 hrs, 1 week, 4 weeks, 6 weeks, 12 weeks
  Early Wound Healing Score (EHS) the following will be assessed and each will be scored from 0 to 2
  1. Clinical signs of re-epithelization (CSR)
  2. Clinical signs of haemostasias (CSH)
  3. Clinical signs of inflammation (CSI)

SECONDARY OUTCOMES:
change in pain scores | 24 hrs, 1 week, 4 weeks
  10-point Visual Analogue Scale (VAS) will be used. A scale of zero to ten (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
change in edema | baseline, 24 hrs, 1 week, 4 weeks, 6 weeks, 12 weeks
  The grading of edema is determined by pit depth (measured visually) and recovery time Ranged from grade 0 (No clinical edema) to grade 4 (Very deep pit (8 mm), more than 30 seconds to rebound)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No